CLINICAL TRIAL: NCT03325517
Title: Effect of Adenovirus E1A Oncogene on DNA Replication Dynamics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Heba Momen kamel (Other)
Responsible Party: Sponsor-Investigator, Heba Momen kamel, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 17200086.
Record Dates: First submitted 2017-10-24; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Adenovirus
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cell lines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND:

The 243 amino acid E1A encoded by the left end of the human adenovirus (Ad) type 2 or 5 genome has been studied in various contexts including as a model cooperating oncoprotein , an apoptosis inducing protein, and as a therapeutic oncolytic protein. All of these properties are associated with its capacity to rapidly induce S phase in a variety of cells. E1A orchestrates most of these effects by interacting with an array of chromatin remodeling complexes, including the Rb family proteins, and the HAT proteins p300 and CBP.

The Myst family protein HBO1 (Myst2, KAT7) is a histone acetyl transferase that plays a major role in replication initiation and also contributes to DNA re-replication. HBO1 directly interacts with Cdt1 and functions as a coactivator of Cdt1 in replication initiation. It also associates with replication origin and stimulates origin activation by acetylating H4 K5, K8, and K12. Overexpression of HBO1 induces DNA re-replication.

SPECIFIC AIM OF THE STUDY: The Specific Aim of this study is to determine whether or not the stimulation of HBO1 activity by E1A plays a role in deregulated DNA replication, and if it does, to determine the mechanism.

1. Using standard assays the investigators will determine whether E1A binds to HBO1 to induce its HAT activity
2. The investigators will determine whether E1A stimulation of HAT activity of HBO1 contributes to DNA re-replication.

RESEARCH DESIGN AND METHODS:

First, the investigators will determine whether E1A associates with replication origins and whether this association requires HBO1. The investigators will use the MCM4 origin which maps in the intergenic region between PRKDC and (Protein Kinase, DNA-Activated, Catalytic Polypeptide) and MCM4 genes.

The investigators will transfect U2OS cells with plasmids expressing relevant proteins then determine their occupancy in origin sequences using ChIP assays. Plasmids expressing epitope tagged WT HBO1 or mutant derivatives along with plasmids expressing WT or mutant E1A proteins will be expressed in U2OS cells, then occupancy of these proteins on origin regions will be quantified using antibodies as appropriate. Typically in these experiments, using relevant antibodies, ChIP assays are performed with primer pairs encompassing origin regions and also regions that are far from origin. Occupancy of initiation factors are increased several fold in the origin region as compared to that of 2KB upstream or downstream regions. Loading of MCM complex along with Cdt1 onto the origins is an indication that initiation of replication occurs in that origin and usually assayed in ChIP-re-ChIP assays as follows: First, loading of HBO1 to the origins will be confirmed using epitope specific antibodies in the first ChIP. The anti-HBO1 precipitates will be re-ChIPed with anti-MCM3 antibodies. Loading of MCM3 helicase to origins occurs after Cdt1 binding and depends on HBO1 HAT activity. Normal amounts of MCM3 will be detected after re-ChIP-ing in E1A+ control samples. If reduced amount of MCM3 is recovered in reChIP assays when mutant E1A or HBO1 mutant (e.g. HBO1 G435A) is used, it would indicate that stimulation of HAT activity by E1A is critical for maximal origin activity in E1A+ cells. This type of assay has considerable flexibility in that mutant proteins can be rapidly assayed. This ChIP-reChiP assays will repeated in different combinations to determine the E1A loading.

These results will be extended to virus infection assays. G1 specific cells isolated by drug treatment will be infected with Ad vectors expressing epitope tagged proteins as appropriate. Association of E1A and HBO1 and their mutant derivatives will be determined. This assay will allow us to confirm the effect of E1A stimulated HAT activity in origin firing and study the effects of E1A on origin firing, if any, other than increasing the HAT activity of HBO1.

DETAILED DESCRIPTION:
BACKGROUND:

TThe 243 amino acid E1A protein (also known as small E1A protein, transforming E1A protein) encoded by the left end of the human adenovirus (Ad) type 2 or 5 genome has been studied in various contexts including as a model cooperating oncoprotein, an apoptosis inducing protein, and as a therapeutic oncolytic protein. All of these properties are associated with its capacity to rapidly induce S phase in a variety of cells. E1A orchestrates most of these effects by interacting with an array of chromatin remodeling complexes, including the Rb family proteins, and the HAT proteins p300 and CBP.

The induction of E2F by E1A-Rb-HDAC interactions is well documented whereas the consequences of E1A-p300/CBP interactions in cell cycle progression are not clear. Previous studies demonstrated that p300/CBP prevents premature entry of quiescent cells into S phase by repressing c-Myc transcription through a tripartite repressor complex consisting of p300, YY1, HDAC3. E1A binds to p300 and dissociates the repressor complex to induce S phase. Induction of c-Myc by this mechanism contributes to the induction of DNA damage response and aberrant cellular DNA replication which leads to genomic instability. In a recently published study, it was shown that E1A induces the pivotal DNA replication initiation factor Cdt1 to high levels resulting in increased replication origin activity and in late S phase, induction of DNA damage response and cellular DNA re-replication. Using the single molecule DNA fiber assay, it was discovered that E1A induces significant changes in the dynamics of DNA replication and appears to induce global changes in origin activation.

Cdt1 is a pivotal DNA replication initiation factor whose levels oscillate during cell cycle progression. In late G1, its levels rise to initiate DNA replication. At the beginning of S phase it is promptly degraded by the E3 ligase so that origins that are already fired once do not fire again in S phase and re-replication within a single cell cycle does not occur. Impaired degradation of Cdt1 in S phase by the E3 ligase is the major mechanism by which the cellular DNA undergoes re-replication. It was discovered that in E1A expressing cells Cdt1 levels remain high in S phase suggesting an inefficient degradation of Cdt1 which may contribute to extensive re-replication of cellular DNA that the investigators observed in late S phase.

The Myst family protein HBO1 (Myst2, KAT7) is a histone acetyl transferase that plays a major role in replication initiation and also contributes to DNA re-replication. HBO1 directly interacts with Cdt1 and functions as a coactivator of Cdt1 in replication initiation. It also associates with replication origin and stimulates origin activation by acetylating H4 K5, K8, and K12. Overexpression of HBO1 induces DNA re-replication. The enrichment of chromatin modifications including acetylation of H4 histones at the origins strongly influences origin activation. Thus, E1A in the absence of a multitude of serum stimulated proliferation signals, forces cells to enter S phase using several compensatory mechanisms. Uncontrolled cellular DNA replication program causes polyploidy that is the hallmark of cancer. It is exciting that a viral oncogene such as E1A alters the cellular DNA replication program. This raises a number of important questions related to the mechanism of replication stress induced by a viral oncogene. For example, how does E1A induce DNA re-replication? Does E1A stimulation of HBO1 alter initiation mechanism and whether HBO1 mediated chromatin modifications at the origins promote re-replication?

SPECIFIC AIM OF THE STUDY:

Our Specific Aim is to determine whether or not the stimulation of HBO1 activity by E1A plays a role in deregulated DNA replication, and if it does, to determine the mechanism.

1. Using standard assays the investigators will determine whether E1A binds to HBO1 to induce its HAT activity
2. Using transient and virus infection assays, the investigators will determine whether stimulation of HBO1 HAT activity by E1A enhances the pre-replicative complex (Pre-RC) formation and whether E1A induced HAT activity qualitatively and quantitatively changes the H4 acetylation at the origin regions.
3. the investigators will determine whether E1A stimulation of HAT activity of HBO1 contributes to DNA re-replication.

RESEARCH DESIGN AND METHODS:

The goal of this study is to determine whether stimulation of HBO1 HAT activity by E1A (i) enhances initiation (ii) induces qualitative and quantitative changes in acetylation of H4 K5, K8 and K12 at the origin region, and (iii) enhances re-replication that occurs in E1A+ cells. If increased HAT activity can stimulate one or more of these functions, it could explain how this property of E1A would contribute to the induction of aberrant DNA replication.

1. E1A binding to WT and HAT deficient HBO1.

   the investigators will first determine whether E1A directly binds to HBO1 by performing the GST binding and in vivo co-IP experiments. If binding is confirmed, the investigators will map the binding sites on both proteins. the investigators will then isolate mutants of both proteins that abolish the interactions. All E1A mutants will be evaluated for their interactions with Rb and p300 and only mutants that retain their capacity to bind to these proteins will be used. It will be necessary to isolate an HBO1 mutant that retains E1A binding capacity but lacks the HAT activity. A widely used HAT deficient mutant G435A will be used in these studies. If E1A binds to this mutant, it will be a valuable mutant to confirm that E1A induced HAT activity is critical for stimulation of replication initiation. If this HBO1 mutant does not bind to E1A, it will be important to isolate new HBO1 mutants which retain E1A binding capacity but lack HAT activity.
2. Role of E1A induced HBO1 HAT activity in origin activation:

   First, the investigators will determine whether E1A associates with replication origins and whether this association requires HBO1. the investigators will use the MCM4 origin which maps in the intergenic region between PRKDC and (Protein Kinase, DNA-Activated, Catalytic Polypeptide) and MCM4 genes. First, the investigators will transfect U2OS cells with plasmids expressing relevant proteins then determine their occupancy in origin sequences using ChIP assays. Plasmids expressing epitope tagged WT HBO1 or mutant derivatives along with plasmids expressing WT or mutant E1A proteins will be expressed in U2OS cells, then occupancy of these proteins on origin regions will be quantified using antibodies as appropriate. Typically in these experiments, using relevant antibodies, ChIP assays are performed with primer pairs encompassing origin regions and also regions that are far from origin. Occupancy of initiation factors are increased several fold in the origin region as compared to that of 2KB upstream or downstream regions. Loading of MCM complex along with Cdt1 onto the origins is an indication that initiation of replication occurs in that origin and usually assayed in ChIP-re-ChIP assays as follows: First, loading of HBO1 to the origins will be confirmed using epitope specific antibodies in the first ChIP. The anti-HBO1 precipitates will be re-ChIPed with anti-MCM3 antibodies. Loading of MCM3 helicase to origins occurs after Cdt1 binding and depends on HBO1 HAT activity. Normal amounts of MCM3 will be detected after re-ChIP-ing in E1A+ control samples. If reduced amount of MCM3 is recovered in reChIP assays when mutant E1A or HBO1 mutant (e.g. HBO1 G435A) is used, it would indicate that stimulation of HAT activity by E1A is critical for maximal origin activity in E1A+ cells. This type of assay which has been successfully used by others has considerable flexibility in that mutant proteins can be rapidly assayed. This ChIP-reChiP assays will repeated in different combinations to determine the E1A loading.

   These results will be extended to virus infection assays. G1 specific cells isolated by drug treatment will be infected with Ad vectors expressing epitope tagged proteins as appropriate. Association of E1A and HBO1 and their mutant derivatives will be determined. This assay will allow us to confirm the effect of E1A stimulated HAT activity in origin firing and study the effects of E1A on origin firing, if any, other than increasing the HAT activity of HBO1. For example, c-Myc induction by E1A does not involve HAT activity.
3. Effects of E1A induced HBO1 HAT activity in the acetylation of H4, K5, K8 and K12.

   To assess this, the investigators will ChIP the chromatin prepared from virus infected cells with the origin specific primers and epitope specific antibodies as appropriate to detect origin loading of HBO1. the investigators will then re-Chip the ChIP precipitates using anti-H4 tetra-Ac antibodies to detect K5, K8, and K12 acetylation. In cells expressing E1A and HBO1, H4 acetylation will be increased considerably as compared to cells infected with HBO1 virus alone. H4 acetylation may be affected depending on the mutants used.
4. E1A stimulated HBO1 HAT activity in re-replication.

   Overexpression of HBO1 has been shown to induce DNA-replication. To determine whether E1A uses HBO1 in inducing re-replication by stimulating the HBO1 HAT activity, the investigators will infect S phase enriched cells (isolated by double thymidine block) with Ad viruses expressing the WT or mutant E1A proteins along with Ad vectors expressing HBO1 variants (e.g. HAT inactive), allow the infection to proceed as needed then quantify the population of cells containing >4N DNA content using flow cytometer. If E1A simulated HBO1 HAT activity is important for re-replication HAT defective HBO1 mutants will not induce re-replication even in the presence of E1A. E1A mutants that cannot bind to HBO1 will also show a similar phenotype.
5. E1A effects on H4 acetylations in re-replicating origins:

   In order to study the H4 acetylations in re-replicating origins, the investigators need to know which of cellular origins undergo re-replication in E1A+ cells in late S phase. the investigators are planning to identify the origins activated in E1A+ cells including those that re-replicate. Once the investigators identify one or two re-replicating origins, the investigators will quantify the acetylations using these origins in cells expressing epitope tagged WT and mutant HBO1 alleles and E1A. the investigators anticipate qualitative or quantitative (or both) in H4 acetylations due to E1A.
6. Expected results and pitfalls:

At the end of all the proposed experiments, the investigators expect to determine whether stimulation of HBO1 HAT activity by E1A is critical for origin activation in E1A+ cells and if E1A induced HAT activity has a role in re-replication. The investigators do not anticipate any technical or other problems including obtaining relevant reagents.

ELIGIBILITY:
Inclusion Criteria:

- All patients who are positive for adenovirus

Exclusion Criteria:

- immune comprised patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are positive for adenovirus (symptomatic or not)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
DNA re-replication indicated by the number of cells containing >4N DNA content using flow cytometer | 1 year
  To determine whether E1A uses HBO1 in inducing re-replication by stimulating the HBO1 HAT activity, the investigators will infect S phase enriched cells (isolated by double thymidine block) with Ad viruses expressing the WT or mutant E1A proteins along with Ad vectors expressing HBO1 variants (e.g. HAT inactive), allow the infection to proceed as needed then quantify the population of cells containing >4N DNA content using flow cytometer. If E1A simulated HBO1 HAT activity is important for re-replication HAT defective HBO1 mutants will not induce re-replication even in the presence of E1A. E1A mutants that cannot bind to HBO1 will also show a similar phenotype.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levine AJ. The common mechanisms of transformation by the small DNA tumor viruses: The inactivation of tumor suppressor gene products: p53. Virology. 2009 Feb 20;384(2):285-93. doi: 10.1016/j.virol.2008.09.034. Epub 2008 Dec 11. PMID 19081592
- [Background] Berk AJ. Recent lessons in gene expression, cell cycle control, and cell biology from adenovirus. Oncogene. 2005 Nov 21;24(52):7673-85. doi: 10.1038/sj.onc.1209040. PMID 16299528
- [Background] DeCaprio JA. How the Rb tumor suppressor structure and function was revealed by the study of Adenovirus and SV40. Virology. 2009 Feb 20;384(2):274-84. doi: 10.1016/j.virol.2008.12.010. Epub 2009 Jan 17. PMID 19150725
- [Background] Breckenridge DG, Shore GC. Regulation of apoptosis by E1A and Myc oncoproteins. Crit Rev Eukaryot Gene Expr. 2000;10(3-4):273-80. doi: 10.1615/critreveukargeneexpr.v10.i3-4.50. PMID 11272469
- [Background] Lavia P, Mileo AM, Giordano A, Paggi MG. Emerging roles of DNA tumor viruses in cell proliferation: new insights into genomic instability. Oncogene. 2003 Sep 29;22(42):6508-16. doi: 10.1038/sj.onc.1206861. PMID 14528275
- [Background] Liao Y, Yu D, Hung MC. Novel approaches for chemosensitization of breast cancer cells: the E1A story. Adv Exp Med Biol. 2007;608:144-69. doi: 10.1007/978-0-387-74039-3_11. PMID 17993239
- [Background] Deissler H, Opalka B. Therapeutic transfer of DNA encoding adenoviral E1A. Recent Pat Anticancer Drug Discov. 2007 Jan;2(1):1-10. doi: 10.2174/157489207779561471. PMID 18221050
- [Background] Smith JG, Wiethoff CM, Stewart PL, Nemerow GR. Adenovirus. Curr Top Microbiol Immunol. 2010;343:195-224. doi: 10.1007/82_2010_16. PMID 20376613
- [Background] Moran E. DNA tumor virus transforming proteins and the cell cycle. Curr Opin Genet Dev. 1993 Feb;3(1):63-70. doi: 10.1016/s0959-437x(05)80342-9. PMID 8453277
- [Background] Kolli S, Buchmann AM, Williams J, Weitzman S, Thimmapaya B. Antisense-mediated depletion of p300 in human cells leads to premature G1 exit and up-regulation of c-MYC. Proc Natl Acad Sci U S A. 2001 Apr 10;98(8):4646-51. doi: 10.1073/pnas.081141998. PMID 11296295
- [Background] Baluchamy S, Rajabi HN, Thimmapaya R, Navaraj A, Thimmapaya B. Repression of c-Myc and inhibition of G1 exit in cells conditionally overexpressing p300 that is not dependent on its histone acetyltransferase activity. Proc Natl Acad Sci U S A. 2003 Aug 5;100(16):9524-9. doi: 10.1073/pnas.1633700100. Epub 2003 Jul 25. PMID 12883011
- [Background] Rajabi HN, Baluchamy S, Kolli S, Nag A, Srinivas R, Raychaudhuri P, Thimmapaya B. Effects of depletion of CREB-binding protein on c-Myc regulation and cell cycle G1-S transition. J Biol Chem. 2005 Jan 7;280(1):361-74. doi: 10.1074/jbc.M408633200. Epub 2004 Nov 2. PMID 15522869
- [Background] Sankar N, Baluchamy S, Kadeppagari RK, Singhal G, Weitzman S, Thimmapaya B. p300 provides a corepressor function by cooperating with YY1 and HDAC3 to repress c-Myc. Oncogene. 2008 Sep 25;27(43):5717-28. doi: 10.1038/onc.2008.181. Epub 2008 Jun 9. PMID 18542060
- [Background] Kadeppagari RK, Sankar N, Thimmapaya B. Adenovirus transforming protein E1A induces c-Myc in quiescent cells by a novel mechanism. J Virol. 2009 May;83(10):4810-22. doi: 10.1128/JVI.02145-08. Epub 2009 Mar 11. PMID 19279113
- [Background] Sankar N, Kadeppagari RK, Thimmapaya B. c-Myc-induced aberrant DNA synthesis and activation of DNA damage response in p300 knockdown cells. J Biol Chem. 2009 May 29;284(22):15193-205. doi: 10.1074/jbc.M900776200. Epub 2009 Mar 30. PMID 19332536
- [Background] Singhal G, Leo E, Setty SK, Pommier Y, Thimmapaya B. Adenovirus E1A oncogene induces rereplication of cellular DNA and alters DNA replication dynamics. J Virol. 2013 Aug;87(15):8767-78. doi: 10.1128/JVI.00879-13. Epub 2013 Jun 5. PMID 23740993
- [Background] Arias EE, Walter JC. Strength in numbers: preventing rereplication via multiple mechanisms in eukaryotic cells. Genes Dev. 2007 Mar 1;21(5):497-518. doi: 10.1101/gad.1508907. PMID 17344412
- [Background] Abbas T, Dutta A. CRL4Cdt2: master coordinator of cell cycle progression and genome stability. Cell Cycle. 2011 Jan 15;10(2):241-9. doi: 10.4161/cc.10.2.14530. Epub 2011 Jan 15. PMID 21212733
- [Background] Avvakumov N, Cote J. Functions of myst family histone acetyltransferases and their link to disease. Subcell Biochem. 2007;41:295-317. PMID 17484133
- [Background] Saksouk N, Avvakumov N, Cote J. (de)MYSTification and INGenuity of tumor suppressors. Cell Mol Life Sci. 2008 Apr;65(7-8):1013-8. doi: 10.1007/s00018-008-7459-x. No abstract available. PMID 18239855
- [Background] Miotto B, Struhl K. HBO1 histone acetylase is a coactivator of the replication licensing factor Cdt1. Genes Dev. 2008 Oct 1;22(19):2633-8. doi: 10.1101/gad.1674108. PMID 18832067
- [Background] Miotto B, Struhl K. HBO1 histone acetylase activity is essential for DNA replication licensing and inhibited by Geminin. Mol Cell. 2010 Jan 15;37(1):57-66. doi: 10.1016/j.molcel.2009.12.012. PMID 20129055
- [Background] Brustel J, Tardat M, Kirsh O, Grimaud C, Julien E. Coupling mitosis to DNA replication: the emerging role of the histone H4-lysine 20 methyltransferase PR-Set7. Trends Cell Biol. 2011 Aug;21(8):452-60. doi: 10.1016/j.tcb.2011.04.006. Epub 2011 May 31. PMID 21632252
- [Background] Vogelauer M, Rubbi L, Lucas I, Brewer BJ, Grunstein M. Histone acetylation regulates the time of replication origin firing. Mol Cell. 2002 Nov;10(5):1223-33. doi: 10.1016/s1097-2765(02)00702-5. PMID 12453428
- [Background] Aggarwal BD, Calvi BR. Chromatin regulates origin activity in Drosophila follicle cells. Nature. 2004 Jul 15;430(6997):372-6. doi: 10.1038/nature02694. PMID 15254542
- [Background] Goren A, Tabib A, Hecht M, Cedar H. DNA replication timing of the human beta-globin domain is controlled by histone modification at the origin. Genes Dev. 2008 May 15;22(10):1319-24. doi: 10.1101/gad.468308. Epub 2008 Apr 28. PMID 18443145
- [Background] Iizuka M, Matsui T, Takisawa H, Smith MM. Regulation of replication licensing by acetyltransferase Hbo1. Mol Cell Biol. 2006 Feb;26(3):1098-108. doi: 10.1128/MCB.26.3.1098-1108.2006. PMID 16428461
- [Background] Abbas T, Shibata E, Park J, Jha S, Karnani N, Dutta A. CRL4(Cdt2) regulates cell proliferation and histone gene expression by targeting PR-Set7/Set8 for degradation. Mol Cell. 2010 Oct 8;40(1):9-21. doi: 10.1016/j.molcel.2010.09.014. PMID 20932471